CLINICAL TRIAL: NCT03857074
Title: Effects of Green Light Exposure on Epileptic Spikes in Patients With Refractory Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alexander Rotenberg, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00030191
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Epilepsy; Epilepsy Intractable
Keywords: Refractory Epilepsy; Green Light Exposure; Epileptic Spikes
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: This is a single-center, open label, pilot feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label, Green Light Exposure (Experimental): This is a single-center, open label, pilot feasibility study. Patients with epilepsy will be exposed to a narrow band of green light at low intensities (1-10 cd/m2). The investigators will record 30 minutes of scalp EEG prior to the light exposure and 30 minutes of scalp EEG recording post-light exposure. The number of epileptic spikes per minute at baseline will be compared to epileptic spike count per minute post-treatment, to determine whether green light exposure effectively decreases the number of epileptic spikes, in patients with ≥1 epileptic spike per minute at baseline.
  Interventions: Device: Green Light Exposure

INTERVENTIONS:
Device: Green Light Exposure — To test whether exposure to a narrow band of green light (520-540 nm) at low intensities (1-10 cd/m2) decreases interictal epileptiform discharges in patients with epilepsy. The overall hypothesis for this open-label trial is based on findings in patients with migraine that indicate an engagement of thalamocortical inhibitory circuits by green light.

SUMMARY:
The purpose of this study is to obtain preliminary data in advance of a larger clinical trial aimed to test whether a single session of green light exposure can lead to a clinically significant reduction in epileptic spikes in patients with medically-refractory epilepsy. As this is a potentially fragile patient population, the study will test safety and tolerability as well as efficacy.

DETAILED DESCRIPTION:
The trial is designed to detect (1) change in spike frequency on EEG before and after exposure to low intensity green light, and (2) presence or absence of neurologic/systemic symptoms referable to exposure of the pre-selected duration, intensity, and band of green light.

Our primary aim is to determine whether prolonged exposure (120 minutes) to a narrow band of green light (520-540 nm) at low intensities (1-10 cd/m2) alters the pattern of electrical activity in the cortex of epilepsy patients.

The primary outcome measure for this aim will be the fraction of patients in which the number of epileptiform discharges (spikes or sharp waves) decrease, per recording, in response to green light exposure, as determined by spike frequency detected via scalp EEG before and after green light exposure.

The investigators anticipate that the primary outcome measures of safety and tolerability will not differ from the previously established measures of green light exposure for migraine (Noseda et al. 2016). The investigators will use only low intensities (1-10 cd/m2) of green light which is well tolerated in adults and children (Main et al. 2000). In addition, given limited experience with conventional green light exposure in epilepsy, the investigators predict that post-exposure to green light, patients will have an improvement on the post-exposure EEG (decreased spike frequency).

ELIGIBILITY:
Inclusion Criteria:

* 6 months-30 years of age
* Epileptic spike frequency ≥1 epileptic spike per minute at baseline, as determined by scalp EEG recording
* Admitted to the Boston Children's Hospital Epilepsy Long Term Monitoring Unit at the time of enrollment

Exclusion Criteria:

* Cataracts
* Retinol disease
* Any history of or currently not well controlled ophthalmic disease that prevents transmission from the retina to the optic nerve
* Clinical seizure 4 hours or less before anticipated green light exposure

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Effects of exposure to a narrow band of green light (520-540 nm) at low intensities (1-10 cd/m2) on the pattern of electrical activity in the cortex of epilepsy patients. | 120 minutes
  The primary outcome measure for this aim will be the fraction of patients in which the number of epileptiform discharges (spikes or sharp waves) decrease, per recording, in response to green light exposure, as determined by spike frequency detected via scalp EEG before and after green light exposure.

SECONDARY OUTCOMES:
To consider probable confounders, such as etiology and comorbidities, this information will be acquired with standardized NIH epilepsy data acquisition forms for (1): | 10 minutes
  Additional anticipated variable (1) patient demographics (age, gender, age of seizure onset, and epilepsy type), will be collected via a 'Demographics' Form.
To consider probable confounders, such as etiology and comorbidities, this information will be acquired through routine clinical care documentation by the study MD for (2): | 10 minutes
  Additional anticipated variable (2) EEG monitoring findings: The study MD will review prior clinical EEG findings per participant.
To consider probable confounders, such as etiology and comorbidities, this information will be acquired through routine clinical care documentation by the study MD for (3): | 10 minutes
  Additional anticipated variable (3) Imaging results: The study MD will review prior clinical imaging findings per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rotenberg, MD, PhD, Principal Investigator — Boston Children's Hospital; Phillip Pearl, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noseda R, Bernstein CA, Nir RR, Lee AJ, Fulton AB, Bertisch SM, Hovaguimian A, Cestari DM, Saavedra-Walker R, Borsook D, Doran BL, Buettner C, Burstein R. Migraine photophobia originating in cone-driven retinal pathways. Brain. 2016 Jul;139(Pt 7):1971-86. doi: 10.1093/brain/aww119. Epub 2016 May 17. PMID 27190022
- [Background] Noseda R, Kainz V, Jakubowski M, Gooley JJ, Saper CB, Digre K, Burstein R. A neural mechanism for exacerbation of headache by light. Nat Neurosci. 2010 Feb;13(2):239-45. doi: 10.1038/nn.2475. Epub 2010 Jan 10. PMID 20062053
- [Background] Noseda R, Lee AJ, Nir RR, Bernstein CA, Kainz VM, Bertisch SM, Buettner C, Borsook D, Burstein R. Neural mechanism for hypothalamic-mediated autonomic responses to light during migraine. Proc Natl Acad Sci U S A. 2017 Jul 11;114(28):E5683-E5692. doi: 10.1073/pnas.1708361114. Epub 2017 Jun 26. PMID 28652355